CLINICAL TRIAL: NCT03141268
Title: Orocecal Transit Time and Fermentation in IBS
Brief Title: Rapid Orocecal Transit Time and Fermentation in IBS.
Acronym: RapidoIBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Per Hellström, Professor, Uppsala University
Other Study IDs: Orocecal lactulose breath
Record Dates: First submitted 2017-04-03; First posted 2017-05-05 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Oro-cecal Transit Time

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: Normal subjects aged 18-80 years. No chronic diseases.
  Interventions: Diagnostic Test: Lactulose breath test
- IBS patients, lactose intolerant: Subjects 18-80 years diagnosed with IBS for more than 6 months ago; lactose intolerant. No concomitant diseases.
  Interventions: Diagnostic Test: Lactulose breath test
- IBS patients, lactose tolerant: Subjects 18-80 years diagnosed with IBS for more than 6 months ago; lactose tolerant. No concomitant diseases.
  Interventions: Diagnostic Test: Lactulose breath test

INTERVENTIONS:
Diagnostic Test: Lactulose breath test — Lactulose 0.67 mg/mL, dose 15 mL (10 grams). No contaminants of lactose. Pharmacy quality.

SUMMARY:
Orocecal transit time is studied in individuals with irritable bowel syndrome (IBS) of both the constipation-dominant, diarrhea-dominant, and mixed form using the lactulose hydrogen breath test for orocecal transit time through the gut. Data are compared to those of healthy volunteers. The peak value of fermentation as read by hydrogen levels is captured after passage of the orocecal segment in the colon. Comparison are made between IBS patients and healthy subjects as regards orocecal transit time and peak fermentation in the cecum.

DETAILED DESCRIPTION:
Patients with IBS of various kind (constipation-dominant, diarrhea-dominant, and mixed form) in large numbers are studied as regards orocecal transit time and compared to healthy controls.

Inclusion criteria: IBS patients 18-80 years old, diagnosis of IBS; exclusion: Severe cardiac, pulmonary, liver or kidney disease, bloody stool After fasting for 12 hours, all subjects ingest 10 grams of lactulose. Hydrogen production, measured as hydrogen concentration in breath, is estimated at 10-minute intervals for a period of 240 minutes. The orocecal transit transit time is measured from ingestion of the lactulose solution until hydrogen peaks to 10 and 20 ppm when passing the ileocecal valve, being fermented by the cecal microflora. Data are compared to those of healthy volunteers.

The peak value of fermentation as read by hydrogen levels (ppm) captured after passage of the ilecocecal valve orocecal valve signifies the gas production of the micro13flora. Comparison are made between IBS patients and healthy subjects as regards orocecal transit time and peak fermentation in the cecum.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, or IBS patients or either kind (IBS-C, IBS-D, IBS-M), no concomitant medication.

Exclusion Criteria:

* Chronic disease, such cardiac, pulmonary, liver, kidney, endocrinological rheumatological, neurological or psychiatric disease plus, in addition, chronic medication.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IBS patients aged 18-80 years of age as recruited in the clinic, some of which are lactose intolerant, others are lactose tolerant.
  Healthy volunteers 18-80 years of age as recruited in society in daily life activities.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Orocecal transit time | 0-240 minutes
  The transit rate of lactulose (foods) through the small intestine

SECONDARY OUTCOMES:
Fermentation of lactulose of the cecal microbiota measured as increase of hydrogen in exhaled breath. | 0-240 minutes
  The rise of hydrogen (beyond 10 and 20 ppm) after lactulose passing the ileo-cecal valve.

CONTACTS AND LOCATIONS:
Overall Officials: Per M Hellstrom, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data are freely available to anyone. Data coded.